CLINICAL TRIAL: NCT06214572
Title: Systemic Therapy With or Without Radiation Therapy in Unresectable Nonmetastatic Gall Bladder Carcinoma: Open Label, Parallel Arm, Phase 2/3 Integrated Randomized Clinical Trial
Brief Title: Radiation Therapy in Unresectable Gall Bladder Cancer
Acronym: RUGB
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Shivakumar Gudi, Assistant Professor, Radiation Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4145
Record Dates: First submitted 2023-12-29; First posted 2024-01-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gall Bladder Cancer
Keywords: Biliary tract cancer; Gall Bladder Cancer; Radiation therapy; Unresectable
MeSH Terms: conditions — Gallbladder Neoplasms; Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; Oxaliplatin; durvalumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systemic therapy (Active Comparator): Participants will receive one of the following Gemcitabine-based systemic therapy alone:
  1. Gemcitabine plus cisplatin:
     Gemcitabine 1000mg/m2 and Cisplatin 25 mg/m2, each administered on Days 1 and 8 every 3 weeks (q3w)
  2. Gemcitabine plus oxaliplatin:
     Gemcitabine 1000 mg/m2 and oxaliplatin 100 mg/m2 IV infusion on days 1 and 8 q2w.
  3. Gemcitabine plus cisplatin plus Durvalumab:
     Durvalumab 1500 mg via intravenous (IV) infusion q4w, starting on Cycle 1 in combination with cisplatin 25 mg/m2 and gemcitabine 1000 mg/m2 each administered on Days 1 and 8, q3w.
  4. Gemcitabine plus cisplatin plus nab-paclitaxel:
  Gemcitabine 800 mg/m2, cisplatin, 25 mg/m2, and nab-paclitaxel 100 mg/m2, on days 1 and 8, q3w.
  duration: 3 months
  Interventions: Drug: Systemic therapy (Gemcitabine plus Cisplatin); Drug: Systemic therapy (Gemcitabine plus oxaliplatin); Drug: Systemic therapy (Gemcitabine plus Cisplatin plus Durvalumab); Drug: Systemic therapy (Gemcitabine plus cisplatin plus nab-paclitaxel)
- RT (Radiation therapy) (Active Comparator): Participants will receive radiation therapy in addition to systemic therapy Hypofractionated external image guided radiation to a dose of 40-55Gy in 10 sessions (up to 60Gy in 15 sessions) over 2-3 weeks.
  This is followed by systemic therapy as in the Systemic therapy arm
  Interventions: Drug: Systemic therapy (Gemcitabine plus Cisplatin); Radiation: RT; Drug: Systemic therapy (Gemcitabine plus oxaliplatin); Drug: Systemic therapy (Gemcitabine plus Cisplatin plus Durvalumab); Drug: Systemic therapy (Gemcitabine plus cisplatin plus nab-paclitaxel)

INTERVENTIONS:
Drug: Systemic therapy (Gemcitabine plus Cisplatin) — Participants will receive one of the following Gemcitabine-based systemic therapy alone:
  Gemcitabine 1000mg/m2 and Cisplatin 25 mg/m2, each administered on Days 1 and 8 every 3 weeks (q3w)
  Duration: 3 months (in addition to 3 months previously received)
Radiation: RT — Participants will receive radiation therapy in addition to systemic therapy Hypofractionated external image guided radiation to a dose of 40-55Gy in 10 sessions (up to 60Gy in 15 sessions) over 2-3 weeks.
  This is followed by systemic therapy as in the Systemic therapy alone arm.
  Arms: RT (Radiation therapy)
Drug: Systemic therapy (Gemcitabine plus oxaliplatin) — Gemcitabine 1000 mg/m2 and oxaliplatin 100 mg/m2 IV infusion on days 1 and 8 q2w.
  Duration: 3 months
Drug: Systemic therapy (Gemcitabine plus Cisplatin plus Durvalumab) — Durvalumab 1500 mg via intravenous (IV) infusion q4w, starting on Cycle 1 in combination with cisplatin 25 mg/m2 and gemcitabine 1000 mg/m2 each administered on Days 1 and 8, q3w.
  Duration 3 months Durvalumab (12 months)
Drug: Systemic therapy (Gemcitabine plus cisplatin plus nab-paclitaxel) — Gemcitabine 800 mg/m2, cisplatin, 25 mg/m2, and nab-paclitaxel 100 mg/m2, on days 1 and 8, q3w Duration: 3 months

SUMMARY:
The goal of this clinical trial is to compare two treatment regimes, namely, systemic therapy (chemotherapy and/or immunotherapy) alone vs. systemic therapy and radiation therapy in patients with inoperable but localized gallbladder cancer. The main questions it aims to answer are:

* Whether adding radiation therapy to systemic therapy improves overall survival?
* What are the effects on other endpoints like cancer-free intervals, side effects, and quality of life? Participants will be randomly assigned to one of the two treatment regimes mentioned earlier by a computer-based program. Researchers will compare survival and quality of life outcomes between the two groups.

DETAILED DESCRIPTION:
Gallbladder cancer (GBC) incidence is exceptionally high in India and most patients present with an unresectable or advanced disease. There is limited clinical evidence on optimal therapy of biliary tract cancers in general and more so for gall bladder cancers which are relatively rare in the Western world.

As per current clinical practice, Surgery remains the mainstay of curative treatment for resectable GBC, and systemic therapy with or without radiotherapy is offered for unresectable GBC. The current standard of systemic therapy is to administer 6 months of Gemcitabine-based regimen and the median overall survival of these patients is about 10-12 months. The national and Institutional guidelines suggest the use of radiation in unresectable GBC. The role of radiation therapy in this setting has not been evaluated in phase 3 randomized clinical trials although it is being offered routinely at our Centre if the patients remain nonmetastatic after initial systemic therapy. We propose a phase 2/3 integrated randomized clinical trial evaluating the role of adding radiotherapy to chemotherapy in improving survival outcomes in patients with unresectable GBC based on nonrandomized data from our institution suggesting a benefit with the addition of radiation therapy in this setting.

Patients with histologically verified, unresectable GBC who do not progress (RECIST 1.1) after an initial 3 months of Gemcitabine-based systemic therapy are invited to participate in this open-label, parallel arm, superiority design randomized controlled trial. Patients randomized to the 'RT arm' will receive hypo fractionated conformal image-guided radiotherapy to a dose of 40-55Gy in 10 (up to 15) fractions to the primary and regional lymph node basins delivered over 2-3 weeks. Systemic therapy is resumed after completion of radiotherapy for 3 more months. The patients in the 'Chemo alone arm' or 'Systemic therapy alone' arm will complete 3 more months of systemic therapy as per the current institutional standard. All patients will be considered for further systemic therapy (either as maintenance therapy or at the time of relapse) at the discretion of the treating medical oncologist.

The primary outcomes of the Phase 2 and Phase 3 components are progression-free survival and Overall survival respectively with an interim analysis planned at 36 months to evaluate futility. Secondary outcomes include local control, toxicity, and quality of life measures. The estimated sample size 249 is and the expected duration of the study is 67 months including the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven (biopsy/cytology) adenocarcinoma of gall bladder. Gall bladder neck primaries with hilar block mimicking hilar cholangiocarcinoma will also be included.
* Non metastatic at presentation as determined using cross sectional imaging and diagnostic laparoscopy if done as a part of standard work up recommended in the joint clinic.
* Locally advanced disease with one or more of the following
* Extensive liver infiltration not amenable for surgery but feasible for safe radiation delivery (Liver minus gross tumor volume at least 700cc)
* Vascular involvement: encasement (>180-degree angle) of one of the vessels: Hepatic artery, main portal vein, right or left portal vein
* Obstructive jaundice with hilar involvement (type 2 non communicating block and higher blocks as per Bismuth-Corlette classification)
* Stable disease or partial response (RECIST 1.1) after initial 3 months of Gemcitabine based chemotherapy
* More than 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 fit for chemotherapy
* Normal hematological and renal and hepatic functions allowing safe delivery of chemotherapy
* Hematological- Hb> 80 g/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L.
* Liver functions- bilirubin ≤ 2 x upper limit normal (ULN), AST/ALT ≤ 5 x ULN, alkaline phosphatase ≤ 6 x upper limit normal (ULN) S. albumin ≥ 30 g/L
* Renal function- Creatinine ≤ 1.5 ULN, Creatinine clearance >= 50 mL/min

Exclusion Criteria:

* Patients with distant metastasis (including nonregional lymph nodes metastasis) will be excluded.
* Prior abdominal therapeutic radiation
* Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
* Pregnancy/Lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2029-07-21 (Estimated); Study Completion 2029-07-21 (Estimated)

PRIMARY OUTCOMES:
Median overall survival | 2 years
  Time interval between the date of diagnosis and death due to any case.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Time interval between the date of diagnosis and radiological or histological (whichever earlier) evidence of disease progression or death from any cause
Locoregional progression free survival | 2 years
  Time interval between the date of diagnosis and radiological or histological (whichever earlier) evidence of locoregional disease progression or death from any cause
Response rate | 6 months
  Response to treatment after completion of 6 months of systemic therapy with or without radiotherapy will be assessed using a PET CT or CECT scan using the RECIST (Ver 1.1) criteria
Acute toxicities | 3 years
  RTOG criteria
Late toxicities | 3 years
  RTOG criteria
Acute toxicities | 3 years
  CTCAE v5 criteria
Late toxicities | 3 years
  CTCAE v5 criteria
Quality of life assessment (Gen) | 2 years
  EORTC QLQ-c30
Quality of life assessment (Liver specific) | 2 years
  FACT-Hep version 4

CONTACTS AND LOCATIONS:
Overall Officials: Shivakumar Gudi, MD, Principal Investigator — Assistant Professor, Radiation Oncology
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma V, Surkar SM, Brooks ED, Simone CB 2nd, Lin C. Chemoradiotherapy Versus Chemotherapy Alone for Unresected Nonmetastatic Gallbladder Cancer: National Practice Patterns and Outcomes. J Natl Compr Canc Netw. 2018 Jan;16(1):59-65. doi: 10.6004/jnccn.2017.7067. PMID 29295882
- [Background] Sinha S, Engineer R, Ostwal V, Ramaswamy A, Chopra S, Shetty N. Radiotherapy for locally advanced unresectable gallbladder cancer - A way forward: Comparative study of chemotherapy versus chemoradiotherapy. J Cancer Res Ther. 2022 Jan-Mar;18(1):147-151. doi: 10.4103/jcrt.JCRT_1568_20. PMID 35381776